CLINICAL TRIAL: NCT04752566
Title: A Phase 3, Prospective, Multicenter, Double Blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of Eculizumab in Patients With Guillain-Barré Syndrome (GBS)
Brief Title: A Study to Evaluate the Efficacy and Safety of Eculizumab in Guillain-Barré Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECU-GBS-301
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Guillain-Barre Syndrome
Keywords: Eculizumab; Soliris; Alexion; C5 Inhibition Therapy
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eculizumab (Experimental): Participants will receive eculizumab.
  Interventions: Biological: Eculizumab
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Eculizumab — Eculizumab will be administered via IV infusion once a week for 4 weeks.
  Other Names: Soliris
  Arms: Eculizumab
Drug: Placebo — Placebo will be administered via IV infusion once a week for 4 weeks.
  Arms: Placebo

SUMMARY:
This is a Phase 3, prospective, multicenter, placebo controlled, double blind, randomized study to investigate the efficacy and safety of eculizumab in participants with severe GBS, defined using the Hughes Functional Grade (FG) scale as progressively deteriorating FG3 or FG4/FG5 within 2 weeks from onset of weakness due to GBS.

This study will be conducted only at sites in Japan.

DETAILED DESCRIPTION:
Eligible participants will be randomized to receive intravenous (IV) infusion of eculizumab or placebo at a 2:1 ratio. All participants will be on concomitant IV immunoglobulin G (Ig) therapy as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the GBS criteria.
* Participants who were able to run prior to onset of GBS symptoms.
* Participants with onset of weakness due to GBS < 2 weeks before screening.
* Participants unable to walk unaided for ≥ 5 meters (progressively deteriorating FG3 or FG4 to FG5).
* Participants who are already on IVIg or deemed eligible for and who will start IVIg.
* Participants who can start their first dose of study drug before the end of the IVIg treatment period.

Exclusion Criteria:

* Participants who have previously received or are currently receiving treatment with complement modulators.
* Participants who have been administered another investigational product within 30 days or 5 half-lives (whichever is longer) prior to providing consent or are currently participating in another interventional study.
* Participants who have received rituximab within 12 weeks prior to screening.
* Participants who are being considered for or are already on plasmapheresis.
* Participants who have received immunosuppressive treatment during the 4 weeks prior to providing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Japan (22):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kagoshima
  - Research Site, Kawagoe-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Kurashiki-shi
  - Research Site, Matsumoto-shi
  - Research Site, Mitaka-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Nishinomiya-shi
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shimotsuga-gun
  - Research Site, Ube-shi
  - Research Site, Yokohama

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were on concomitant intravenous immunoglobulin (IVIg) therapy as per standard of care.
Groups:
- Eculizumab: Participants received eculizumab intravenous (IV) infusion on Days 1, 8, 15, and 22.
- Placebo: Participants received placebo matched to eculizumab via IV infusion on Days 1, 8, 15, and 22.
Period: Overall Study
Arm/Group | Eculizumab | Placebo
Started | 37 | 20
Received at Least 1 Dose of Study Drug | 37 | 20
Completed | 32 | 18
Not Completed | 5 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had a baseline functional grade (FG) score and at least 1 postbaseline FG score.
Groups:
- Eculizumab: Participants received eculizumab IV infusion on Days 1, 8, 15, and 22.
- Total: Total of all reporting groups
Arm/Group | Eculizumab | Placebo | Total
Number analyzed (Participants) | 37 | 20 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (19.61) | 56.2 (18.34) | 56.4 (19.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 24
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 20 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 20 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Reaching a Hughes Functional Grade (FG) Score <=1
Description: The mobility of the participants was evaluated on a 7 point disability functional grade scale and described as Hughes FG score of 0 (Healthy, no signs or symptoms of Guillain-Barré syndrome); 1 (Minor signs or symptoms and able to run); 2 (Able to walk 5 metre (m) across an open space without assistance); 3 (Able to walk 5 m across an open space with the help of one person and waist-level walking-frame, stick, or sticks); 4 (Chairbound/bedbound: unable to walk as in 3); 5 (Requiring assisted ventilation [for at least part of day or night]) and 6 (Dead), where higher numbers indicate more severe impairment. The Kaplan-Meier estimate of time to event of FG<=1 is reported. Time (days) to first event=Date of first event-Date of first dose+1. Participants who discontinued early without achieving FG <= 1 were censored at the date of discontinuation. Participants who completed the study without achieving FG<=1 were censored at the date of study completion.
Time Frame: Up to Week 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had a baseline FG score and at least 1 postbaseline FG score. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 20 | 13
Days | 112.0 [59.0 to NA] — NA signifies upper limit was not estimable as study does not have enough events to estimate the median time to event. | 168.0 [36.0 to NA] — NA signifies upper limit was not estimable as study does not have enough events to estimate the median time to event.
Statistical Analysis 1: Comparison: Eculizumab vs Placebo; Test type: Superiority; p = 0.8938, Log Rank — Log Rank Test stratified by randomization strata; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.45 to 1.97] — Cox proportional hazard model stratified by randomization strata, with treatment group as the fixed effect. Firth's adjustment was applied if no event was observed in a treatment group

2. Secondary Outcome: Number of Participants With A Hughes Functional Grade (FG) Score <=1
Description: The mobility of the participants was evaluated on a 7 point disability FG scale and described as Hughes FG score of 0 (Healthy, no signs or symptoms of Guillain-Barré syndrome); 1 (Minor signs or symptoms and able to run); 2 (Able to walk 5 m across an open space without assistance); 3 (Able to walk 5 m across an open space with the help of one person and waist-level walking-frame, stick, or sticks); 4 (Chairbound/bedbound: unable to walk as in 3); 5 (Requiring assisted ventilation [for at least part of day or night]) and 6 (Dead), where higher numbers indicate more severe impairment. If a participant had an FG score <= 1 prior to or at Week 8 and Week 24, respectively, then the participant is considered a responder. Otherwise, participants discontinued prior to Week 8 and Week 24 or with an FG score > 1 at Week 8 and Week 24 are nonresponders, respectively.
Time Frame: Week 8, Week 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had a baseline FG score and at least 1 postbaseline FG score.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 37 | 20
Participants
  Week 8 | 12 | 7
  Week 24 | 20 | 13
Statistical Analysis 1: Comparison: Eculizumab vs Placebo; Week 8; Test type: Superiority; p = 0.8987, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.27 to 3.17]
Statistical Analysis 2: Comparison: Eculizumab vs Placebo; Week 24; Test type: Superiority; p = 0.4083, Regression, Logistic; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.18 to 2.02]

3. Secondary Outcome: Number of Participants With A Hughes Functional Grade Score Improvement of >=3
Description: The mobility of the participants was evaluated on a 7 point disability FG scale and described as Hughes FG score of 0 (Healthy, no signs or symptoms of Guillain-Barré syndrome); 1 (Minor signs or symptoms and able to run); 2 (Able to walk 5 m across an open space without assistance); 3 (Able to walk 5 m across an open space with the help of one person and waist-level walking-frame, stick, or sticks); 4 (Chairbound/bedbound: unable to walk as in 3); 5 (Requiring assisted ventilation [for at least part of day or night]) and 6 (Dead), where higher numbers indicate more severe impairment. Participants with a change from baseline in FG score (value at Week 24 - baseline value) <= -3 were considered a responder. Participants with change from baseline > -3 and participants who discontinued prior to Week 24 were considered non-responders.
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 37 | 20
Participants | 16 | 10
Statistical Analysis 1: Comparison: Eculizumab vs Placebo; Test type: Superiority; p = 0.6739, Regression, Logistic; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.24 to 2.54]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as an adverse event (AE) with onset on or after the first dose of the study drug. An AE is any untoward medical occurrence in a participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 up to Week 24
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 37 | 20
Participants | 34 | 19

5. Secondary Outcome: Free Complement Component 5 in Serum
Time Frame: Week 24
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study drug and who have at least 1 postdose PD sample. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 32 | 18
micrograms/milliliters | 131.0438 (29.40068) | 147.8833 (36.70182)

6. Secondary Outcome: Hemolytic Complement Activity in Serum
Time Frame: Week 24
Population: Pharmacodynamic analysis set included all participants who received at least 1 dose of study drug and who have at least 1 postdose PD sample. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of hemolysis
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 32 | 18
percentage of hemolysis | 91.79 (11.077) | 91.83 (11.767)

7. Secondary Outcome: Length of Stay in the Hospital
Description: For participants with multiple hospitalizations, the total duration of all hospitalizations was summarized.
Time Frame: Up to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 37 | 20
days | 49.5 (27.15) | 39.8 (12.97)

8. Secondary Outcome: Number of Participants Who Required Mechanical Ventilator Support
Description: For participants with more than 1 episode of the same support, the total duration across all episodes was summarized.
Time Frame: Up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 37 | 20
Participants | 8 | 1

9. Secondary Outcome: Concentration of Eculizumab in Serum
Time Frame: Up to Week 24
Population: Pharmacokinetic analysis set (PKAS) included all participants who received at least 1 dose of study drug and who had at least 1 postdose PK sample. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters
Arm/Group | Eculizumab
Number analyzed (Participants) | 32
micrograms/milliliters | 4.690 (0.0000)

10. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies
Time Frame: Up to Week 12
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 37 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 24
Description: Safety set included all participants who received at least 1 dose of study drug.
Arm/Group | Eculizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/37 | 1/20
Other Adverse Events (participants affected / at risk) | 34/37 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=37) | Placebo (N=20)
Hanging (General disorders) | 1 | 0
Pneumonia aspiration (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=37) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Dry eye (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 5 | 0
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 3
Pneumonia aspiration (Infections and infestations) | 5 | 2
COVID-19 (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Genital candidiasis (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3
Alanine aminotransferase increased (Investigations) | 1 | 3
Liver function test increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Protein urine (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 10 | 8
Delirium (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 1
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT04752566/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT04752566/SAP_001.pdf